CLINICAL TRIAL: NCT03861572
Title: Eccentric Training Effects on Functionality and on Triceps Surae Neuromechanical Properties After Achilles Tendon Surgical Repair
Brief Title: Eccentric Training Effects on Functionality and Neuromechanical Properties After Achilles Tendon Surgical Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Marco Aurélio Vaz, PhD, Principal Investigator, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFRGS 3.046.049
Record Dates: First submitted 2019-02-25; First posted 2019-03-04 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Achilles Tendon Rupture
Keywords: Achilles tendon; physical therapy; eccentric training; Achilles tendon rupture; rehabilitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Raters will be blinded to the participants' allocation in each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isokinetic eccentric group (Experimental): The isokinetic eccentric training will be carried out with the volunteers positioned seated on the dynamometer with the apparent axis of the ankle joint rotation aligned with the dynamometer's axis of rotation. Movement will be executed in the angular velocity of 30°·s-1. Ankle range of motion (ROM) will be standardized for all participants in 50º, which shall respect each individual's maximal dorsiflexion amplitude. The 50° eccentric training ROM will start from each subject's 80% of the maximal dorsiflexion. This procedure will be used to ensure that all subjects perform training on the same plantar flexor muscular length, which should promote the same level of muscular requirement among the participants. This methodology was recently used by GEREMIA and VAZ (2016) study.
  Interventions: Other: Isokinetic eccentric training
- Traditional eccentric training (Active Comparator): Participants will be engaged in an intervention program consisting of 12 weeks of traditional eccentric training. The training will be carried out with the volunteers at gym in stand position. Concentric phase will be realized with both legs and the eccentric one only with one of them. Training progression will be the same from de isokinetic eccentric group. The same periodization from eccentric group will be used to permit us a posteriori comparison between groups. Training sessions will be performed at university gym, twice a week, with a minimum interval of 72 hours between sessions. Each training session will comprise the same specific warming protocol for the ankle joint from the eccentric training.
  Interventions: Other: Traditional eccentric training

INTERVENTIONS:
Other: Isokinetic eccentric training — Training sessions will be performed in the same isokinetic dynamometer used in previous evaluations, twice a week, with a minimum interval of 72 hours between sessions.
  Arms: Isokinetic eccentric group
Other: Traditional eccentric training — Training sessions will be performed at university gym, twice a week, with a minimum interval of 72 hours between sessions.
  Arms: Traditional eccentric training

SUMMARY:
Early rehabilitation protocols have been studied in Achilles tendon (AT) rupture patients, but deficits in tendon biomechanical properties have been observed several years after the injury. AT rupture patients are unable to return to their previous levels of physical activity. They present deleterious adaptations in the plantar flexor muscles that lead to functional deficits, and deficits in the tendon's structural and mechanical properties. Eccentric contractions have been suggested to recover these muscle properties. This contraction is known to produce higher force compared to isometric and concentric contractions, and increases tendon stiffness. However, there is a lack of studies showing the effects of the eccentric training in AT rupture rehabilitation. We want to know if an isokinetic eccentric training program will determine the desired adaptations on triceps surae muscle-tendon unit's properties in patients subjected to the AT surgical repair. More specifically, the aim of this study is verifying the effects of a 12-week eccentric training program on triceps surae muscle-tendon unit's properties in subjects that were subjected to the AT surgical repair. 30 subjects will be randomized in two groups: (1) isokinetic eccentric training; and (2) traditional eccentric training control group. All participants will be submitted to a four-week control period, followed by a 12-week period of training for the plantar flexor muscles. Neuromuscular system properties, AT biomechanical properties and functional tests will be evaluated. Participants will be evaluated in four moments: at baseline; after 4, 8 and 12 weeks of rehabilitation. Tendon mechanical (stiffness, stress, strain), material (Young's modulus) and morphological (cross-sectional area and tendon length) properties; muscle architecture (thickness, pennation angle and fascicle length); and functional tests (heel rise resistance and height) will be analyzed between groups and periods. Effects and interactions will be analyzed with ANOVA two-way. Clinical effects will be analyzed using effect size and magnitude-based inferences.

DETAILED DESCRIPTION:
Detailed Description: Early rehabilitation protocols have been studied in Achilles tendon (AT) rupture patients, but deficits in tendon biomechanical properties have been observed several years after the injury. AT rupture patients are unable to return to their previous levels of physical activity. They present deleterious adaptations in the plantar flexor muscles that lead to functional deficits and deficits in the tendon structural and mechanical properties. Deficits in calf muscle endurance and strength remained 7 years after the injury. In this regards, eccentric contractions are recommended to recover muscle morphology and mechanical properties. This contraction type produces higher force compared to isometric and concentric contractions, and increases tendon stiffness. However, there is a lack of studies showing the effect of the eccentric training in AT rupture rehabilitation. We want to know if an isokinetic eccentric training program will determine the desired adaptations on triceps surae muscle-tendon unit's properties in patients subjected to the AT surgical repair. More specifically, the aim of this study is verifying the effects of a 12-week eccentric training program on triceps surae muscle-tendon unit's properties in subjects that were subjected to the AT surgical repair. Our hypothesis is that the eccentric training program will (1) increase the ability to produce muscular strength; (2) will produce an increase in gastrocnemius and soleus muscles thickness, fascicle length, and pennation angle; (3) will increase AT stiffness and Young's modulus; (4) will increase ankle functionality; (5) will improve the patient's quality of life. Finally, we expect that the abovementioned changes from isokinetic eccentric training will be greater than those from the traditional eccentric control group that will be subjected to 12 weeks of plantar flexor training with weights. 30 subjects will be randomized in two groups: (1) isokinetic eccentric training; and (2) traditional eccentric training control group. All participants will be submitted to a four-week control period, followed by a 12- week period of training for the plantar flexor muscles. Neuromuscular system properties, AT biomechanical properties and functional tests will be evaluated. Participants will be evaluated in four moments: at baseline; after 4, 8 and 12 weeks of rehabilitation. Tendon mechanical (stiffness, stress, strain), material (Young's modulus) and morphological (cross sectional area and tendon length) properties; muscle architecture (thickness, pennation angle and fascicle length); and functional tests (heel rise resistance and height) will be analyzed between groups and periods. Effects and interactions will be analyzed with ANOVA two- way (group x period). Clinical effects will be analyzed using effect size (Cohen's d) and magnitude-based inferences.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be male and female subjects who suffered total acute Achilles tendon rupture, and which underwent surgical repair. In addition, to participate in this study all volunteers will need to present medical and/or physiotherapeutic release for physical/sports activities practice.

Exclusion Criteria:

* Volunteers that did not have Achilles tendon surgical reconstruction, that did not present medical and/or physiotherapeutic release for physical/sports activities, who have participated in strength training program for the plantar flexors in the last 6 months, patients with diabetic diseases, as well as those with difficulty for understanding and/or executing the test and training protocols in the isokinetic dynamometer will be excluded.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Tendon Young's modulus | First evaluation, change from baseline to 4 weeks of training, change from baseline to 8 weeks of training and change from baseline to 12 weeks of training
  Tendon elastic modulus (Young's modulus) will be obtained by calculating the slope in the last 40% of the linear region of the stress-strain curve.
Tendon stiffness | First evaluation, change from baseline to 4 weeks of training, change from baseline to 8 weeks of training and change from baseline to 12 weeks of training
  Tendon stiffness will be obtained by calculating the slope in the last 40% of the linear region of the force-deformation curve.
Resistance to plantar flexion test | First baseline evaluation, change from baseline to 4 weeks of training, change from baseline to 8 weeks of training and change from baseline to 12 weeks of training
  The number of times, as well as the elevation height, will be used for data analysis. Height will be recorded and will be analyzed with Kinovea software.
Vertical countermovement jump | First baseline evaluation, change from baseline to 4 weeks of training, change from baseline to 8 weeks of training and change from baseline to 12 weeks of training
  Vertical jump will be recorded using cameras and maximal vertical height will be measured using Kinovea software.
Triple hop test | First baseline evaluation, change from baseline to 4 weeks of training, change from baseline to 8 weeks of training and change from baseline to 12 weeks of training
  Maximal distance of a triple unilateral jump will be measure with a metric tape.

SECONDARY OUTCOMES:
Achilles tendon cross-sectional area | First evaluation, change from baseline to 4 weeks of training, change from baseline to 8 weeks of training and change from baseline to 12 weeks of training
  To obtain the Achilles tendon cross-sectional area (CSA), the US probe (GE Healthcare, Waukesha, Washington, USA) will be placed perpendicular to the tendon (in the transverse plane), and 3 images will be obtained with reference to the distances of 2, 4, 6, 8 and 10 cm of the muscle insertion in the calcaneus bone (ARYA and KULIG, 2010). Area values will be obtained for each image, and the final value of the area will be calculated by the average of these five values.
Achilles tendon length | First evaluation, change from baseline to 4 weeks of training, change from baseline to 8 weeks of training and change from baseline to 12 weeks of training
  To obtain Achilles tendon length, the US (LOGIQ P6, GE Healthcare, Waukesha, Washington, USA) and a linear matrix array transducer (GE Healthcare, Waukesha, Washington, USA) will be placed longitudinally to the tendon (in the sagittal plane). The most distal portion of the Achilles tendon, inserted into the calcaneus bone, will be determined by US, and the respective point will be marked on the skin. After this, the probe will be moved to a proximal position until the visualization of the medial gastrocnemius myotendinous junction (MTJ), which is also marked on the skin. The distance between the two marked points on the skin will be measured with a measuring tape, this distance being considered representative of the tendon length (ARYA and KULIG, 2010; GEREMIA et al., 2015; GEREMIA and VAZ, 2016).
Muscle strength | First evaluation, change from baseline to 4 weeks of training, change from baseline to 8 weeks of training and change from baseline to 12 weeks of training
  The plantar flexor capacity of force production will be obtained during isometric and isokinetic tests using an isokinetic dynamometer (Biodex System 3 Pro, Biodex Medical Systems, USA). Firstly, the isometric tests will be performed, followed by the concentric and eccentric tests.
Muscle Architecture | First evaluation, change from baseline to 4 weeks of training, change from baseline to 8 weeks of training and change from baseline to 12 weeks of training
  Muscular architecture will be evaluated with an US system and a linear matrix array probe (GE Healthcare, Waukesha, Washington, USA). Muscle architecture parameters will involve fascicle length, pennation angle and muscle thickness (NARICI, 1999). Echo-intensity of the medial gastrocnemius will also be evaluated. The images will be obtained with the subjects in the ventral decubitus position on a stretcher, with the knees extended and the ankle in neutral position (heel line at a 90° angle with respect to the longitudinal axis of the leg, 0° of plantarflexion). A custom system will be used to secure the ankle in the neutral position. The probe will be positioned longitudinally to the muscle fibers at 30% proximal for medial and lateral gastrocnemius, and 50% for soleus, of the distance between the popliteal fold and the lateral malleolus center (KAWAKAMI et al., 1998).
Resistance to plantar flexion test | First evaluation, change from baseline to 4 weeks of training, change from baseline to 8 weeks of training and change from baseline to 12 weeks of training
  The number of times, as well as the elevation height, will be used for data analysis.
Calf muscle perimetry | First evaluation, change from baseline to 4 weeks of training, change from baseline to 8 weeks of training and change from baseline to 12 weeks of training
  To calculate the calf muscles perimetry, the leg length will be determined from the distance between the center of the lateral malleolus and the popliteal fossa at the knee. From the determination of this distance, the value corresponding to 30% of the distance from the articular line of the knee will be calculated for the measurement of the leg perimetry (MIYATANI et al., 2004)
Muscle echo-intensity | First evaluation, change from baseline to 4 weeks of training, change from baseline to 8 weeks of training and change from baseline to 12 weeks of training
  For the echo-intensity evaluation, the probe will be positioned transversally at the proximal 30% of the lower leg length (AKAGI et al., 2018). Three images will be recorded in the same position of the muscle architecture. Echo-intensity has been associated with force production (CADORE et al., 2012; RECH et al., 2014; AKAGI et al., 2018), an aspect that we want to analyze is if there is some correlation among structural and functional variables
Muscle Activation | First evaluation, change from baseline to 4 weeks of training, change from baseline to 8 weeks of training and change from baseline to 12 weeks of training
  Gastrocnemius and sóleo muscles electromyography (EMG) signals will be measured through pairs of passive surface electrodes (Ag/AgCl, Meditrace, Kendall, Canada) in bipolar configuration. A reference electrode will be placed on the skin covering the anterior surface of the tibia, according to the procedures proposed by the Surface Electromyography for the Non-Invasive Assessment of Muscles (SENIAM, 2018). The electrodes will be fixed on the skin and a slight pressure will be applied on them to increase the contact between the electrode gel and the skin. The electrodes placement will respect the recommendations proposed by (SENIAM, 2018).

CONTACTS AND LOCATIONS:
Overall Officials: Marco A Vaz, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Exercise Research Laboratory, School of Physical Education, Physical Therapy and Dance, Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Barfod KW, Hansen MS, Holmich P, Troelsen A, Kristensen MT. Efficacy of early controlled motion of the ankle compared with no motion after non-operative treatment of an acute Achilles tendon rupture: study protocol for a randomized controlled trial. Trials. 2016 Nov 29;17(1):564. doi: 10.1186/s13063-016-1697-2. PMID 27894329
- [Background] Baroni BM, Geremia JM, Rodrigues R, De Azevedo Franke R, Karamanidis K, Vaz MA. Muscle architecture adaptations to knee extensor eccentric training: rectus femoris vs. vastus lateralis. Muscle Nerve. 2013 Oct;48(4):498-506. doi: 10.1002/mus.23785. Epub 2013 Jul 15. PMID 23852989
- [Background] Baroni BM, Rodrigues R, Franke RA, Geremia JM, Rassier DE, Vaz MA. Time course of neuromuscular adaptations to knee extensor eccentric training. Int J Sports Med. 2013 Oct;34(10):904-11. doi: 10.1055/s-0032-1333263. Epub 2013 Mar 22. PMID 23526592
- [Background] Batterham AM, Hopkins WG. Making meaningful inferences about magnitudes. Int J Sports Physiol Perform. 2006 Mar;1(1):50-7. PMID 19114737
- [Background] BENJAMIN, M.; THEOBALD, P.; SUZUKI, D. et al. The Anatomy of the Achilles Tendon. In: MAFFULLI, N. e ALMEKINDERS, L. C. (Ed.). The Achilles Tendon. London, UK: Springer, 2007. cap. 2,
- [Background] Brorsson A, Gravare Silbernagel K, Olsson N, Nilsson Helander K. Calf Muscle Performance Deficits Remain 7 Years After an Achilles Tendon Rupture. Am J Sports Med. 2018 Feb;46(2):470-477. doi: 10.1177/0363546517737055. Epub 2017 Oct 25. PMID 29068725
- [Background] Brorsson A, Willy RW, Tranberg R, Gravare Silbernagel K. Heel-Rise Height Deficit 1 Year After Achilles Tendon Rupture Relates to Changes in Ankle Biomechanics 6 Years After Injury. Am J Sports Med. 2017 Nov;45(13):3060-3068. doi: 10.1177/0363546517717698. Epub 2017 Aug 7. PMID 28783473
- [Background] Chalmers J. Review article: Treatment of Achilles tendon ruptures. J Orthop Surg (Hong Kong). 2000 Jun;8(1):97-99. doi: 10.1177/230949900000800118. No abstract available. PMID 12468884
- [Background] COHEN, J. Statistical Power Analysis for the Behavioral Sciences. 2nd. USA: Lawrence Erlbaum Associates, Publishers, 1988.
- [Background] Duclay J, Martin A, Duclay A, Cometti G, Pousson M. Behavior of fascicles and the myotendinous junction of human medial gastrocnemius following eccentric strength training. Muscle Nerve. 2009 Jun;39(6):819-27. doi: 10.1002/mus.21297. PMID 19301364
- [Background] El-Akkawi AI, Joanroy R, Barfod KW, Kallemose T, Kristensen SS, Viberg B. Effect of Early Versus Late Weightbearing in Conservatively Treated Acute Achilles Tendon Rupture: A Meta-Analysis. J Foot Ankle Surg. 2018 Mar-Apr;57(2):346-352. doi: 10.1053/j.jfas.2017.06.006. Epub 2017 Sep 30. PMID 28974345
- [Background] Frankewycz B, Krutsch W, Weber J, Ernstberger A, Nerlich M, Pfeifer CG. Rehabilitation of Achilles tendon ruptures: is early functional rehabilitation daily routine? Arch Orthop Trauma Surg. 2017 Mar;137(3):333-340. doi: 10.1007/s00402-017-2627-9. Epub 2017 Jan 17. PMID 28097423
- [Background] Frizziero A, Trainito S, Oliva F, Nicoli Aldini N, Masiero S, Maffulli N. The role of eccentric exercise in sport injuries rehabilitation. Br Med Bull. 2014 Jun;110(1):47-75. doi: 10.1093/bmb/ldu006. Epub 2014 Apr 15. PMID 24736013
- [Background] Frizziero A, Vittadini F, Fusco A, Giombini A, Masiero S. Efficacy of eccentric exercise in lower limb tendinopathies in athletes. J Sports Med Phys Fitness. 2016 Nov;56(11):1352-1358. Epub 2015 Nov 26. PMID 26609968
- [Background] Geremia JM, Bobbert MF, Casa Nova M, Ott RD, Lemos Fde A, Lupion Rde O, Frasson VB, Vaz MA. The structural and mechanical properties of the Achilles tendon 2 years after surgical repair. Clin Biomech (Bristol). 2015 Jun;30(5):485-92. doi: 10.1016/j.clinbiomech.2015.03.005. Epub 2015 Mar 11. PMID 25828432
- [Background] Gomes da Silva CF, Lima E Silva FX, Vianna KB, Oliveira GDS, Vaz MA, Baroni BM. Eccentric training combined to neuromuscular electrical stimulation is not superior to eccentric training alone for quadriceps strengthening in healthy subjects: a randomized controlled trial. Braz J Phys Ther. 2018 Nov-Dec;22(6):502-511. doi: 10.1016/j.bjpt.2018.03.006. Epub 2018 Mar 28. PMID 29628406
- [Background] Heikkinen J, Lantto I, Piilonen J, Flinkkila T, Ohtonen P, Siira P, Laine V, Niinimaki J, Pajala A, Leppilahti J. Tendon Length, Calf Muscle Atrophy, and Strength Deficit After Acute Achilles Tendon Rupture: Long-Term Follow-up of Patients in a Previous Study. J Bone Joint Surg Am. 2017 Sep 20;99(18):1509-1515. doi: 10.2106/JBJS.16.01491. PMID 28926379
- [Background] Herzog W, ter Keurs HE. Force-length relation of in-vivo human rectus femoris muscles. Pflugers Arch. 1988 Jun;411(6):642-7. doi: 10.1007/BF00580860. PMID 3412867
- [Background] Horstmann T, Lukas C, Merk J, Brauner T, Mundermann A. Deficits 10-years after Achilles tendon repair. Int J Sports Med. 2012 Jun;33(6):474-9. doi: 10.1055/s-0032-1301932. Epub 2012 Apr 12. PMID 22499571
- [Background] Huang J, Wang C, Ma X, Wang X, Zhang C, Chen L. Rehabilitation regimen after surgical treatment of acute Achilles tendon ruptures: a systematic review with meta-analysis. Am J Sports Med. 2015 Apr;43(4):1008-16. doi: 10.1177/0363546514531014. Epub 2014 May 2. PMID 24793572
- [Background] Karamanidis K, Arampatzis A. Mechanical and morphological properties of human quadriceps femoris and triceps surae muscle-tendon unit in relation to aging and running. J Biomech. 2006;39(3):406-17. doi: 10.1016/j.jbiomech.2004.12.017. PMID 16389081
- [Background] Korkmaz M, Erkoc MF, Yolcu S, Balbaloglu O, Oztemur Z, Karaaslan F. Weight bearing the same day versus non-weight bearing for 4 weeks in Achilles tendon rupture. J Orthop Sci. 2015 May;20(3):513-6. doi: 10.1007/s00776-015-0710-z. Epub 2015 Mar 14. PMID 25773309
- [Background] Langberg H, Ellingsgaard H, Madsen T, Jansson J, Magnusson SP, Aagaard P, Kjaer M. Eccentric rehabilitation exercise increases peritendinous type I collagen synthesis in humans with Achilles tendinosis. Scand J Med Sci Sports. 2007 Feb;17(1):61-6. doi: 10.1111/j.1600-0838.2006.00522.x. Epub 2006 Jun 19. PMID 16787448
- [Background] Lantto I, Heikkinen J, Flinkkila T, Ohtonen P, Kangas J, Siira P, Leppilahti J. Early functional treatment versus cast immobilization in tension after achilles rupture repair: results of a prospective randomized trial with 10 or more years of follow-up. Am J Sports Med. 2015 Sep;43(9):2302-9. doi: 10.1177/0363546515591267. Epub 2015 Jul 30. PMID 26229048
- [Background] Lantto I, Heikkinen J, Flinkkila T, Ohtonen P, Leppilahti J. Epidemiology of Achilles tendon ruptures: increasing incidence over a 33-year period. Scand J Med Sci Sports. 2015 Feb;25(1):e133-8. doi: 10.1111/sms.12253. Epub 2014 May 23. PMID 24862178
- [Background] MAFFULLI, N.; ALMEKINDERS, L. C. The Achilles Tendon. Springer, 2007.
- [Background] Maffulli N, Tallon C, Wong J, Lim KP, Bleakney R. Early weightbearing and ankle mobilization after open repair of acute midsubstance tears of the achilles tendon. Am J Sports Med. 2003 Sep-Oct;31(5):692-700. doi: 10.1177/03635465030310051001. PMID 12975188
- [Background] Maffulli N, Walley G, Sayana MK, Longo UG, Denaro V. Eccentric calf muscle training in athletic patients with Achilles tendinopathy. Disabil Rehabil. 2008;30(20-22):1677-84. doi: 10.1080/09638280701786427. PMID 18608370
- [Background] Mahieu NN, McNair P, Cools A, D'Haen C, Vandermeulen K, Witvrouw E. Effect of eccentric training on the plantar flexor muscle-tendon tissue properties. Med Sci Sports Exerc. 2008 Jan;40(1):117-23. doi: 10.1249/mss.0b013e3181599254. PMID 18091014
- [Background] McNair P, Nordez A, Olds M, Young SW, Cornu C. Biomechanical properties of the plantar flexor muscle-tendon complex 6 months post-rupture of the Achilles tendon. J Orthop Res. 2013 Sep;31(9):1469-74. doi: 10.1002/jor.22381. Epub 2013 May 6. PMID 23649780
- [Background] Morrissey D, Roskilly A, Twycross-Lewis R, Isinkaye T, Screen H, Woledge R, Bader D. The effect of eccentric and concentric calf muscle training on Achilles tendon stiffness. Clin Rehabil. 2011 Mar;25(3):238-47. doi: 10.1177/0269215510382600. Epub 2010 Oct 27. PMID 20980351
- [Background] Mortensen HM, Skov O, Jensen PE. Early motion of the ankle after operative treatment of a rupture of the Achilles tendon. A prospective, randomized clinical and radiographic study. J Bone Joint Surg Am. 1999 Jul;81(7):983-90. doi: 10.2106/00004623-199907000-00011. PMID 10428130
- [Background] Neumayer F, Mouhsine E, Arlettaz Y, Gremion G, Wettstein M, Crevoisier X. A new conservative-dynamic treatment for the acute ruptured Achilles tendon. Arch Orthop Trauma Surg. 2010 Mar;130(3):363-8. doi: 10.1007/s00402-009-0865-1. Epub 2009 Apr 2. PMID 19340434
- [Background] Pensini M, Martin A, Maffiuletti NA. Central versus peripheral adaptations following eccentric resistance training. Int J Sports Med. 2002 Nov;23(8):567-74. doi: 10.1055/s-2002-35558. PMID 12439772
- [Background] Valkering KP, Aufwerber S, Ranuccio F, Lunini E, Edman G, Ackermann PW. Functional weight-bearing mobilization after Achilles tendon rupture enhances early healing response: a single-blinded randomized controlled trial. Knee Surg Sports Traumatol Arthrosc. 2017 Jun;25(6):1807-1816. doi: 10.1007/s00167-016-4270-3. Epub 2016 Aug 18. PMID 27539402
- [Background] Wasielewski NJ, Kotsko KM. Does eccentric exercise reduce pain and improve strength in physically active adults with symptomatic lower extremity tendinosis? A systematic review. J Athl Train. 2007 Jul-Sep;42(3):409-21. PMID 18059998
- [Background] Zellers JA, Carmont MR, Gravare Silbernagel K. Return to play post-Achilles tendon rupture: a systematic review and meta-analysis of rate and measures of return to play. Br J Sports Med. 2016 Nov;50(21):1325-1332. doi: 10.1136/bjsports-2016-096106. Epub 2016 Jun 3. PMID 27259751
- [Background] Zhang H, Tang H, He Q, Wei Q, Tong D, Wang C, Wu D, Wang G, Zhang X, Ding W, Li D, Ding C, Liu K, Ji F. Surgical Versus Conservative Intervention for Acute Achilles Tendon Rupture: A PRISMA-Compliant Systematic Review of Overlapping Meta-Analyses. Medicine (Baltimore). 2015 Nov;94(45):e1951. doi: 10.1097/MD.0000000000001951. PMID 26559266